CLINICAL TRIAL: NCT02525458
Title: Antimicrobial Activity of a Quaternary Ammonium Methacryloxy Silicate-containing Acrylic Resin: A Randomized Clinical Trial
Brief Title: Quaternary Ammonium Methacryloxy Silicate-containing Acrylic Resin
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Frank Tay, BDSc (Hons), PhD (Other)
Collaborators: Wuhan University (Other); Washington University School of Medicine (Other); Air Force Military Medical University, China (Other); Tongji Hospital (Other); Augusta University (Other)
Responsible Party: Sponsor-Investigator, Frank Tay, BDSc (Hons), PhD, Doctor, Kimmerling Holdings Group, LLC
Organization: Kimmerling Holdings Group, LLC (Other)
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Supportive Care
Other Study IDs: QAMS-2015
Record Dates: First submitted 2015-08-09; First posted 2015-08-17 (Estimated); Last update posted 2016-08-30 (Estimated); Status verified 2016-08

CONDITIONS: Oral Health
Keywords: antimicrobial; biofilms; acrylic resin; polymethyl methacrylate; confocal laser scanning microscopy; split-mouth design; quaternary ammonium methacryloxy silicate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- QAMS-containing PMMA (Experimental): PMMA containing 5% QAMS
  Interventions: Device: QAMS-containing PMMA
- QAMS-free PMMA (Placebo Comparator): PMMA containing 0% QAMS
  Interventions: Device: QAMS-free PMMA

INTERVENTIONS:
Device: QAMS-containing PMMA — Wear retainer with QMAS-containing PMMA on one side of retainer
  Arms: QAMS-containing PMMA
Device: QAMS-free PMMA — Wear retainer with QMAS-free PMMA on other side of retainer
  Arms: QAMS-free PMMA

SUMMARY:
One of the major challenges in orthodontic treatment is long-term stability. Because removable retainers are worn for at least one year, bacteria and fungi may accumulate on the retainers in the form of multi-species plaque biofilms. This may result in increased incidence of proximal dental caries or oral candida infection. Thus, incorporation of antimicrobial activity in orthodontic acrylic resin to achieve plaque biofilm reduction is highly desirable. An antimicrobial and antifungal quaternary ammonium methacryloxy silicate molecule (QAMS) has been synthesized by sol-gel reaction and incorporated into orthodontic acrylic resin. The QAMS-copolymerized acrylic resin demonstrated contact-killing properties against single-species biofilms in previous in vitro studies and has received US FDA 510(K) clearance for marketing. The objective of the present randomized clinical trial is to determine the in vivo antimicrobial efficacy of the QAMS-containing orthodontic acrylic by using removable retainers that are worn by recruited subjects to create 48-hour multi-species plaque biofilms. The null hypothesis tested is that there is no difference in the antimicrobial activities between QAMS-free and QAMS-containing orthodontic acrylic resin on oral biofilms grown in vivo in human subjects.

DETAILED DESCRIPTION:
There is increasing demand for orthodontic care worldwide. In the United States, approximately one-fifth of the adolescents and teenagers, and up to 1% of young adults are receiving some form of the orthodontic treatment. One of the major challenges in orthodontic treatment is long-term stability; removable and fixed retainers are required to stabilise the aligned dentition and prevent post-treatment relapse. Most removable retainers are constructed of polymethyl methacrylates (PMMA), which are held by metal clasps around the posterior teeth. Because removable retainers are worn in a moist intraoral environment with fluctuating pH for at least one year, bacteria and fungi may accumulate on or within the retainers in the form of multi-species plaque biofilms that act as reservoirs of these microorganisms. This may result in increased incidence of proximal dental caries or oral candidiasis. Moreover, other opportunistic pathogens such as methicillin-resistant Staphylococcus aureus have been identified from orthodontic retainers, which may potentially lead to local or systemic infection, particularly in orthodontic patients with complicated medical disorders. For adult patients, oral microorganisms derived from removable acrylic appliances have been implicated in bacteria endocarditis, pneumonia, chronic obstructive pulmonary disease and gastrointestinal infection. Production of volatile odoriferous compounds by colonized microorganisms also contributes to halitosis, which affects a person's communication and psychological well-being.

Microbial plaque biofilm accumulation on removable orthodontic appliances and retainers is usually controlled by mechanical and chemical means. Despite their effectiveness, these procedures demand stringent patient compliance, which may not be readily achievable in those with restricted dexterity. Hence, incorporation of antimicrobial activity in orthodontic acrylic resin to achieve plaque biofilm reduction is highly desirable. Conventional PMMA-based antimicrobial approaches are based on leaching of antimicrobial agents of small molecular mass (e.g. chlorhexidine) into the intraoral environment, application of an antimicrobial coating on the surface of the material or incorporation of antibacterial silver nanoparticles into the PMMA resin. Antimicrobial polymers are rapidly becoming a new class of biomaterials that can be functionalized and tethered to materials and kill microbes without releasing the biocides. For methacrylates, anionic and phosphated PMMA polymers have been created that can copolymerize with PMMA to create acrylic resins with permanent, non-leaching antimicrobial properties.

Cationic polymers containing quaternary ammonium and phosphonium groups possess contact-killing antimicrobial activities. An antimicrobial and antifungal cationic quaternary ammonium methacryloxy silicate molecule (QAMS) has been synthesized by sol-gel reaction between a tetraalkoxysilane and two trialkoxysilanes. Containing a methacryloxy functional group and a long C-18 carbon chain, the QAMS molecule is soluble in MMA monomer and has been incorporated into PMMA orthodontic acrylic resin. The QAMS-copolymerised acrylic resin demonstrated improved fracture toughness without adversely affecting flexural modulus and strength of the orthodontic acrylic. In previous in vitro studies, orthodontic acrylic resins containing 4-6% QAMS were found to possess in vitro immediate diffusional as well as contact-killing antimicrobial properties when tested with Streptococcus mutans, Actinomyces naeslundii and Candida albicans. To investigate the antimicrobial durability of the QAMS-containing acrylic resin, specimens were aged in water for 3 months prior to evaluation of their antimicrobial activities. Even after 3 months of water-ageing wherein any residual effects of diffusional kill would have been completely eliminated, the QAMS-containing orthodontic acrylic resin still possessed antimicrobial activities against single-species biofilms generated from the three microbes. Antimicrobial polymers designed for biomedical applications should also be minimally cytotoxic to host tissues. In a previous study, the viability of an odontoblast-like cell line derived from mouse dental papilla was examined by exposing these cells to QAMS-containing orthodontic acrylic resin. Results of the cell viability assays indicated that the QAMS-containing orthodontic acrylic resin is relatively non-cytotoxic. The QAMS-containing orthodontic acrylic has received 510(K) clearance for marketing by the U.S. Food and Drug Administration (FDA). Nevertheless, clinical trials are lacking that demonstrate the in vivo antimicrobial potential of QAMS-containing orthodontic acrylic on multi-species biofilms.

Although various multi-species oral biofilm models have been developed and have contributed to the understanding of intraoral microbial adhesion and biofilm formation, these models have drawbacks in that they are unlikely to replicate the variability and in vivo dynamics of plaque biofilms. Apart from differences in structural characteristics between in vitro and in vivo biofilms, the presence of host defenses such as antimicrobial peptides derived from saliva, is seldom take into account in in vitro multi-species biofilm models. More than 600 microbial species have been identified in the human oral microflora, of which approximately 280 species have been isolated in culture. Thus, plaque biofilm profiles are unique among individuals, being modulated by different environmental factors as well as variable quorum sensing signals derived from adjacent microorganisms. These confounding factors may temper the efficacy of antimicrobial polymers in vivo. Accordingly, the objective of the present randomised clinical trial was to determine the in vivo antimicrobial efficacy of the FDA-approved QAMS-containing orthodontic acrylic by using custom-made removable Hawley retainers that were worn intraorally by recruited subjects to create 48-hour multi-species plaque biofilms. Because of the anticipated high variability in the microbial composition of individual plaque biofilms, a split-mouth design was utilised to reduce inter-subject variability, with procedures taken to minimize unwanted carry-across effects. The null hypothesis tested was that there is no difference in the antimicrobial activities between QAMS-free and QAMS-containing orthodontic acrylic resin on oral biofilms grown in vivo in human subjects.

ELIGIBILITY:
Inclusion Criteria:

* Healthy individual with no history or presence of a systemic disease
* Absence of active caries or periodontal disease with pocket depths deeper than 4 mm

Exclusion Criteria:

* Extensive gag reflex that precludes taking of an intraoral alginate impression
* Presence of cleft palate that precludes the wearing of a Hawley retainer
* Have been using an antimicrobial mouthwash prior to enrolment in the study
* Have been taking antibiotics against infectious diseases in the half year preceding the study

Ages: 21 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2015-07; Primary Completion 2015-10 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
Biofilm killing efficacy within the biovolume (3D) and biomass (2D) of multi-species biofilms measured by confocal laser scanning microscopy and image analysis | 48 hours
  Percentage kill of microorganisms ranging from 0% (no kill) to 100% (complete eradication of microorganisms within biofilm)

SECONDARY OUTCOMES:
Redness, inflammation, ulceration or swelling of oral mucosa | 48 hours
  Adverse effects in the form of redness, inflammation, ulceration or swelling of oral mucosa

CONTACTS AND LOCATIONS:
Overall Officials: Siying Liu, PhD, Study Director — School & Hospital of Stomatology, Wuhan University
Locations (1):
- School and Hospital of Stomatology, Wuhan University, Wuhan, Hubei, China

REFERENCES:
- [Background] Okunseri C, Pajewski NM, McGinley EL, Hoffmann RG. Racial/ethnic disparities in self-reported pediatric orthodontic visits in the United States. J Public Health Dent. 2007 Fall;67(4):217-23. doi: 10.1111/j.1752-7325.2007.00032.x. PMID 18087992
- [Background] Whitesides J, Pajewski NM, Bradley TG, Iacopino AM, Okunseri C. Socio-demographics of adult orthodontic visits in the United States. Am J Orthod Dentofacial Orthop. 2008 Apr;133(4):489.e9-14. doi: 10.1016/j.ajodo.2007.08.016. PMID 18405809
- [Background] Littlewood SJ, Millett DT, Doubleday B, Bearn DR, Worthington HV. Orthodontic retention: a systematic review. J Orthod. 2006 Sep;33(3):205-12. doi: 10.1179/146531205225021624. PMID 16926314
- [Background] Pathak AK, Sharma DS. Biofilm associated microorganisms on removable oral orthodontic appliances in children in the mixed dentition. J Clin Pediatr Dent. 2013 Spring;37(3):335-9. doi: 10.17796/jcpd.37.3.92230h6256v8697t. PMID 23855182
- [Background] Batoni G, Pardini M, Giannotti A, Ota F, Giuca MR, Gabriele M, Campa M, Senesi S. Effect of removable orthodontic appliances on oral colonisation by mutans streptococci in children. Eur J Oral Sci. 2001 Dec;109(6):388-92. doi: 10.1034/j.1600-0722.2001.00089.x. PMID 11767275
- [Background] Addy M, Shaw WC, Hansford P, Hopkins M. The effect of orthodontic appliances on the distribution of Candida and plaque in adolescents. Br J Orthod. 1982 Jul;9(3):158-63. doi: 10.1179/bjo.9.3.158. PMID 6954991
- [Background] Bjerklin K, Garskog B, Ronnerman A. Proximal caries increment in connection with orthodontic treatment with removable appliances. Br J Orthod. 1983 Jan;10(1):21-4. doi: 10.1179/bjo.10.1.21. PMID 6573195
- [Background] Hibino K, Wong RW, Hagg U, Samaranayake LP. The effects of orthodontic appliances on Candida in the human mouth. Int J Paediatr Dent. 2009 Sep;19(5):301-8. doi: 10.1111/j.1365-263X.2009.00988.x. Epub 2009 Apr 16. PMID 19486368
- [Background] Chang CS, Al-Awadi S, Ready D, Noar J. An assessment of the effectiveness of mechanical and chemical cleaning of Essix orthodontic retainer. J Orthod. 2014 Jun;41(2):110-7. doi: 10.1179/1465313313Y.0000000088. Epub 2014 Feb 17. PMID 24536071
- [Background] Patel A, Burden DJ, Sandler J. Medical disorders and orthodontics. J Orthod. 2009 Dec;36 Suppl:1-21. doi: 10.1179/14653120723346. PMID 19934236
- [Background] Coulthwaite L, Verran J. Potential pathogenic aspects of denture plaque. Br J Biomed Sci. 2007;64(4):180-9. doi: 10.1080/09674845.2007.11732784. PMID 18236742
- [Background] Verran J. Malodour in denture wearers: an ill-defined problem. Oral Dis. 2005;11 Suppl 1:24-8. doi: 10.1111/j.1601-0825.2005.01083.x. PMID 15752093
- [Background] Vento-Zahra E, De Wever B, Decelis S, Mallia K, Camilleri S. Randomized, double-blind, placebo-controlled trial to test the efficacy of nitradine tablets in maxillary removable orthodontic appliance patients. Quintessence Int. 2011 Jan;42(1):37-43. PMID 21206932
- [Background] Fathi H, Martiny H, Jost-Brinkmann PG. Efficacy of cleaning tablets for removable orthodontic appliances: an in vivo pilot study. J Orofac Orthop. 2015 Mar;76(2):143-51. doi: 10.1007/s00056-014-0277-x. English, German. PMID 25746845
- [Background] Kenawy el-R, Worley SD, Broughton R. The chemistry and applications of antimicrobial polymers: a state-of-the-art review. Biomacromolecules. 2007 May;8(5):1359-84. doi: 10.1021/bm061150q. Epub 2007 Apr 11. PMID 17425365
- [Background] Raj PA, Dentino AR. Denture polymers with antimicrobial properties: a review of the development and current status of anionic poly(methyl methacrylate) polymers. Future Med Chem. 2013 Sep;5(14):1635-45. doi: 10.4155/fmc.13.145. PMID 24047269
- [Background] Carmona-Ribeiro AM, de Melo Carrasco LD. Cationic antimicrobial polymers and their assemblies. Int J Mol Sci. 2013 May 10;14(5):9906-46. doi: 10.3390/ijms14059906. PMID 23665898
- [Background] Gong SQ, Niu LN, Kemp LK, Yiu CK, Ryou H, Qi YP, Blizzard JD, Nikonov S, Brackett MG, Messer RL, Wu CD, Mao J, Bryan Brister L, Rueggeberg FA, Arola DD, Pashley DH, Tay FR. Quaternary ammonium silane-functionalized, methacrylate resin composition with antimicrobial activities and self-repair potential. Acta Biomater. 2012 Sep;8(9):3270-82. doi: 10.1016/j.actbio.2012.05.031. Epub 2012 May 29. PMID 22659173
- [Background] Gong SQ, Epasinghe J, Rueggeberg FA, Niu LN, Mettenberg D, Yiu CK, Blizzard JD, Wu CD, Mao J, Drisko CL, Pashley DH, Tay FR. An ORMOSIL-containing orthodontic acrylic resin with concomitant improvements in antimicrobial and fracture toughness properties. PLoS One. 2012;7(8):e42355. doi: 10.1371/journal.pone.0042355. Epub 2012 Aug 1. PMID 22870322
- [Background] Gong SQ, Epasinghe DJ, Zhou B, Niu LN, Kimmerling KA, Rueggeberg FA, Yiu CK, Mao J, Pashley DH, Tay FR. Effect of water-aging on the antimicrobial activities of an ORMOSIL-containing orthodontic acrylic resin. Acta Biomater. 2013 Jun;9(6):6964-73. doi: 10.1016/j.actbio.2013.02.031. Epub 2013 Feb 26. PMID 23485857
- [Background] Shu M, Wong L, Miller JH, Sissons CH. Development of multi-species consortia biofilms of oral bacteria as an enamel and root caries model system. Arch Oral Biol. 2000 Jan;45(1):27-40. doi: 10.1016/s0003-9969(99)00111-9. PMID 10669090
- [Background] Guggenheim B, Guggenheim M, Gmur R, Giertsen E, Thurnheer T. Application of the Zurich biofilm model to problems of cariology. Caries Res. 2004 May-Jun;38(3):212-22. doi: 10.1159/000077757. PMID 15153691
- [Background] Chavez de Paz LE. Development of a multispecies biofilm community by four root canal bacteria. J Endod. 2012 Mar;38(3):318-23. doi: 10.1016/j.joen.2011.11.008. Epub 2012 Jan 5. PMID 22341068
- [Background] Al-Ahmad A, Wunder A, Auschill TM, Follo M, Braun G, Hellwig E, Arweiler NB. The in vivo dynamics of Streptococcus spp., Actinomyces naeslundii, Fusobacterium nucleatum and Veillonella spp. in dental plaque biofilm as analysed by five-colour multiplex fluorescence in situ hybridization. J Med Microbiol. 2007 May;56(Pt 5):681-687. doi: 10.1099/jmm.0.47094-0. PMID 17446294
- [Background] Zijnge V, van Leeuwen MB, Degener JE, Abbas F, Thurnheer T, Gmur R, Harmsen HJ. Oral biofilm architecture on natural teeth. PLoS One. 2010 Feb 24;5(2):e9321. doi: 10.1371/journal.pone.0009321. PMID 20195365
- [Background] van 't Hof W, Veerman EC, Nieuw Amerongen AV, Ligtenberg AJ. Antimicrobial defense systems in saliva. Monogr Oral Sci. 2014;24:40-51. doi: 10.1159/000358783. Epub 2014 May 23. PMID 24862593
- [Background] Bjarnsholt T, Alhede M, Alhede M, Eickhardt-Sorensen SR, Moser C, Kuhl M, Jensen PO, Hoiby N. The in vivo biofilm. Trends Microbiol. 2013 Sep;21(9):466-74. doi: 10.1016/j.tim.2013.06.002. Epub 2013 Jul 2. PMID 23827084
- [Background] Dewhirst FE, Chen T, Izard J, Paster BJ, Tanner AC, Yu WH, Lakshmanan A, Wade WG. The human oral microbiome. J Bacteriol. 2010 Oct;192(19):5002-17. doi: 10.1128/JB.00542-10. Epub 2010 Jul 23. PMID 20656903
- [Background] Toyofuku M, Inaba T, Kiyokawa T, Obana N, Yawata Y, Nomura N. Environmental factors that shape biofilm formation. Biosci Biotechnol Biochem. 2016;80(1):7-12. doi: 10.1080/09168451.2015.1058701. Epub 2015 Jun 23. PMID 26103134
- [Background] Dixon EF, Hall RA. Noisy neighbourhoods: quorum sensing in fungal-polymicrobial infections. Cell Microbiol. 2015 Oct;17(10):1431-41. doi: 10.1111/cmi.12490. Epub 2015 Sep 3. PMID 26243526
- [Background] Lesaffre E, Philstrom B, Needleman I, Worthington H. The design and analysis of split-mouth studies: what statisticians and clinicians should know. Stat Med. 2009 Dec 10;28(28):3470-82. doi: 10.1002/sim.3634. PMID 19536744
- [Background] Pandis N, Walsh T, Polychronopoulou A, Katsaros C, Eliades T. Split-mouth designs in orthodontics: an overview with applications to orthodontic clinical trials. Eur J Orthod. 2013 Dec;35(6):783-9. doi: 10.1093/ejo/cjs108. Epub 2013 Feb 1. PMID 23376899
- See also: Statistical Brief #368. Agency for Healthcare Research and Quality, Rockville, MD. — http://meps.ahrq.gov/mepsweb/data_files/publications/st368/stat368.shtml
- See also: 25. U. S. Food and Drug Administration. 510(k) premarket notification — http://www.accessdata.fda.gov/scripts/cdrh/cfdocs/cfpmn/pmn.cfm?ID=K141439